CLINICAL TRIAL: NCT02059980
Title: Developing Effective Response Inhibition Training for Symptom Relief in Obsessive-Compulsive and Related Disorders and Trichotillomania
Brief Title: Developing Effective Response Inhibition Training for Symptom Relief in OCD and Trichotillomania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Han Joo Lee, Assistant Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21-RIT_OC-LEE; R21MH094537 (NIH)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Obsessive Compulsive Disorder; Trichotillomania
Keywords: OCD; Trichotillomania; Response inhibition; Cognitive training
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Trichotillomania

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Response inhibition training (Experimental): Eight 45-minute sessions of computerized training on response inhibition over a 4 week period
  Interventions: Behavioral: Response inhibition training
- Placebo Control Training (Placebo Comparator): Eight 45-minute sessions of computerized placebo control training over a 4 week period
  Interventions: Behavioral: Placebo Control Training

INTERVENTIONS:
Behavioral: Response inhibition training — This is a computerized video game that offers 40 training levels, which aims to enhance the individual's response inhibition performance
  Arms: Response inhibition training
Behavioral: Placebo Control Training — This placebo control training looks very similar to the response inhibition training program in its appearance. However, it does not offer any practice related to response inhibition capabilities.
  Arms: Placebo Control Training

SUMMARY:
Obsessive-compulsive disorder (OCD) and its related disorders (e.g., trichotillomania) are characterized by the marked difficulty in inhibiting unwanted or inappropriate responses. There is compelling evidence that poor response inhibition is a core cognitive feature of OCD and its related disorders, but no effective intervention exists that directly attempts to address this problematic cognitive deficiency. This study will examine the feasibility and clinical utility of a computerized cognitive training program designed to improve response inhibition among individuals diagnosed with OCD or trichotillomania.This training program offers systematic practice of response inhibition in the form of a 40-level computer game. Individuals with these conditions will be randomized to either 8 sessions of (a) computerized response inhibition training (RIT) or (b) placebo computer training (PLT). We hypothesize that RIT will outperform PLT in improving response inhibition capabilities and reducing relevant clinical symptoms. In sum, this project is expected to generate important knowledge to guide the development of effective computer-based treatment approaches that may help reduce critical problems of existing treatments such as suboptimal patient retention and treatment under-utilization, thereby improving overall treatment response rates among individuals suffering from OCD and related conditions.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of obsessive-compulsive disorder or trichotillomania

Exclusion Criteria:

* Current substance use problems
* Current/Past Psychotic disorder, bipolar disorder, or schizophrenia
* Attention deficit/hyperactivity disorder or tic disorder
* Severe depressive symptoms
* Current psychotherapy
* Current suicidality
* Estimated intellectual functioning < 80
* Lack of response inhibition deficits on a stop-signal task

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Joo Lee, Ph.D., Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- Psychology Clinic, University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled individuals diagnosed with obsessive-compulsive disorder or trichotillomania at a mid-west university in the United States. The last participant completed in August 2017.
Pre-assignment Details: For this study, 258 individuals underwent online pre-screenings, and 83 participated in onsite full eligibility assessments. A total of 45 individuals met the study entry criteria, and were invited to the main study. Of them, 33 participants completed pre-training assessment and randomized into one of the two training conditions.
Period: Overall Study
Arm/Group | Response Inhibition Training | Placebo Control Training
Started | 18 | 15
Completed | 16 | 14
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Response Inhibition Training | Placebo Control Training | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.17 (12.01) | 24.47 (5.48) | 28.67 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 14 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 14 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 15 | 33
Depression Anxiety and Stress - 21 [Mean (Standard Deviation); unit: units on a scale] — The Depression Anxiety and Stress - 21 (DASS21) is a widely used questionnaire for assessment general emotional distress, including depression, anxiety, and stress symptoms. We examined the total score on the measure (range: 0 ~ 63), with the higher scores indicating a greater level of emotional distress.
  units on a scale | 27.56 (24.08) | 29.73 (17.00) | 28.55 (20.88)
Obsessive-Compulsive Inventory-Revised [Mean (Standard Deviation); unit: units on a scale] — The Obsessive-Compulsive Inventory-Revised (OCI-R) is a widely used self-report measure for assessing symptoms of OCD. The possible range of the total scores is 0 ~ 72. The table reports the total scores on the OCI-R, with higher scores indicating a greater level of OCD symptom severity.
  units on a scale | 20.61 (16.96) | 19.60 (12.57) | 20.15 (14.91)

OUTCOME MEASURES:

1. Primary Outcome: Composite Score of Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) and National Institute of Mental Health (NIMH)
Description: This is a clinician-administered rating scale of OCD symptom severity, most widely used in treatment outcome research for OCD, and a clinician-administered rating scale of hair pulling symptoms, widely used in clinical trial research for trichotillomania. Given the inclusion of two different diagnostic conditions, the primary outcome for the current study is the z score of the symptom rating severity obtained from the two rating scales, with higher values indicating greater symptom severity.
Time Frame: Baseline, Week 4, and Week 8
Population: Intent to treat population (all participants who received at least one session of training with a pre-training assessment). Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: z scores
Arm/Group | Response Inhibition Training | Placebo Control Training
Number analyzed (Participants) | 18 | 15
z scores
  Baseline | -.38 (1.13) | .46 (.51)
  Week 4 | -.89 (1.83) | -.52 (1.20)
  Week 8 | -1.20 (2.03) | -.71 (1.68)
Statistical Analysis 1: Comparison: Response Inhibition Training vs Placebo Control Training; It was calculated that 30 participants rnadomized in a 1:1 fashion between the 2 arms would have .90 power to detect a large effect (f=.40), but is somewhat underpowered to detect a medium effect (f=.25) between the two groups. Sample size was determined using a repeated-measures ANOVA test (α = .05, a correlation of .5 among repeated measures, and a nonsphericity correction of .6), considering the design effect and potential patient attrition (=25%); Test type: Superiority; p = 0.56, Mixed Models Analysis

2. Primary Outcome: Stop Signal Reaction Time
Description: Stop Signal Reaction Time (SSRT; time taken to complete the inhibitory process) is estimated using the tracking algorithm on the computerized stop-signal task, which adjusts the stop signal delay automatically (by 50ms) to maintain the rate of successful inhibition on stop-signal trials at 50%.
Time Frame: Baseline, Week 4, and Week 8
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Response Inhibition Training | Placebo Control Training
Number analyzed (Participants) | 18 | 15
milliseconds
  Baseline | 225.47 (29.10) | 225.83 (18.96)
  Week 4 | 215.68 (21.74) | 212.92 (18.82)
  Week 8 | 211.46 (21.99) | 208.69 (42.77)
Statistical Analysis 1: Comparison: Response Inhibition Training vs Placebo Control Training; It was calculated that 30 participants randomized in a 1:1 fashion between the 2 arms would have .90 power to detect a large effect (f=.40), but is somewhat underpowered to detect a medium effect (f=.25) between the two groups. Sample size was determined using a repeated-measures ANOVA test (α = .05, a correlation of .5 among repeated measures, and a nonsphericity correction of .6), considering the design effect and potential patient attrition (=25%); Test type: Superiority; p = .98, Mixed Models Analysis

3. Secondary Outcome: Clinical Global Impression Severity and Improvement
Description: The Clinical Global Impression Severity and Improvement (CGI) is a clinician-administered rating scale widely used to assess the overall severity of the target condition in treatment outcome research. The CGI is assessed on a 7-point scale, with the severity scale from 1 (Normal, not at all ill) through to 7 (Among the most severely ill patients). Thus, the higher CGI severity rating score indicate a greater level of overall illness.
Time Frame: Baseline, Week 4, and Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Response Inhibition Training | Placebo Control Training
Number analyzed (Participants) | 18 | 15
score on a scale
  Baseline | 3.67 (.69) | 4.00 (.54)
  Week 4 | 3.63 (.89) | 3.57 (.65)
  Week 8 | 3.20 (1.01) | 3.69 (.75)

4. Secondary Outcome: Commission Errors on the Go/No-go Task.
Description: The number of commission errors on the go/no-go task is a commonly used measure of response inhibition. In this task, participants are asked to withhold their responses on no-go trials. If they fail to withhold their response in a no-go trial (i.e., pressing the response key to the no-go signal), this response counts toward the total number of commission errors. Therefore, a greater number of commission errors on this task reflects a greater level of inhibitory control deficit.
Time Frame: Baseline, Week 4, and Week 8
Measure: Mean (Standard Deviation); unit: The number of commission errors
Arm/Group | Response Inhibition Training | Placebo Control Training
Number analyzed (Participants) | 18 | 15
The number of commission errors
  Baseline | 10.41 (6.76) | 9.40 (5.78)
  Week 4 | 10.69 (5.75) | 15.64 (8.90)
  Week 8 | 9.38 (4.32) | 11.77 (7.24)

ADVERSE EVENTS:
Time Frame: The occurrence of adverse events were collected throughout the main assessment time points, including baseline, post-training, and 1-month follow-up assessments. Thus, the time window has been about 2 months for participants.
Arm/Group | Response Inhibition Training | Placebo Control Training
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 0/18 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02059980/Prot_SAP_000.pdf